CLINICAL TRIAL: NCT02369341
Title: A Phase III Study for the Evaluation of the Immunogenicity and Reactogenicity of GSK Biologicals' Quadrivalent Split Virion Influenza Vaccine Fluarix Tetra (2015 Season Southern Hemisphere) in Adults 18 Years of Age and Above
Brief Title: Immunogenicity and Reactogenicity of GlaxoSmithKline (GSK) Biologicals' Quadrivalent Split Virion Influenza Vaccine Fluarix Tetra (2015 Season Southern Hemisphere) in Adults 18 Years of Age and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201959
Record Dates: First submitted 2015-02-16; First posted 2015-02-23 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-09

CONDITIONS: Influenza
Keywords: Southern Hemisphere influenza vaccine; Elderly; Seasonal flu; Fluarix Tetra; Adults; Immunogenicity; Reactogenicity; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluarix Tetra (Southern Hemisphere) Adult Group (Experimental): Subjects aged 18-60 years received 1 dose of Fluarix™ Tetra (Southern Hemisphere) vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: Fluarix Tetra
- Fluarix Tetra (Southern Hemisphere) Elderly Group (Experimental): Subjects aged >60 years received 1 dose of Fluarix™ Tetra (Southern Hemisphere) vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: Fluarix Tetra

INTERVENTIONS:
Biological: Fluarix Tetra — One dose of the Fluarix™ Tetra vaccine was administered to all subjects on Day 0 (Visit 1) intramuscularly into the deltoid of the non-dominant arm.
  Other Names: FLU D-QIV (GSK Biologicals' Quadrivalent Split Virion Influenza Vaccine Fluarix Tetra); Influsplit™ Tetra

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of GSK Biologicals' Quadrivalent Split Virion Influenza Vaccine Fluarix Tetra (2015 Southern hemisphere) in adults (18 to 60 years of age) and in the elderly (over 60 years of age).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing any study specific procedure.
* A male or female aged 18 years or above at the time of vaccination.
* Healthy subjects with well-controlled chronic diseases as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine during the period starting 30 days before the dose of study vaccine (Day -29 to Day 0), or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the vaccine dose. For corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs (e.g. rituximab, infliximab, etc.) within 6 months before study start, or planned administration during the study.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the study vaccination and during the entire study period.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the first dose of study vaccine or planned administration during the study period.
* Administration of an influenza vaccine within the 6 months preceding the study start or planned use of such vaccines during the study period..
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Clinically or virologically confirmed influenza infection within the six months preceding the study vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 38.0°C/100.4°F, measured by any means.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Chronic underlying disease (such as cancer, chronic obstructive pulmonary disease under oxygen therapy, insulin-dependent diabetes mellitus), not stabilised or clinically serious.
* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* History of Guillain-Barré syndrome.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine, including latex.
* History of severe adverse reaction to a previous influenza vaccination.
* Anaphylaxis following the administration of vaccine(s).
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2015-06-03 (Actual); Study Completion 2015-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Brazil (2):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 201959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was allocated the subject number but did not receive the study vaccination.
Period: Overall Study
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Started | 63 | 57
Completed | 62 | 57
Not Completed | 1 | 0
Not completed — Migrated/moved from study area | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group | Total
Number analyzed (Participants) | 63 | 57 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.8 (12.2) | 67.2 (6.0) | 53.3 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 38 | 90
  Male | 11 | 19 | 30

OUTCOME MEASURES:

1. Primary Outcome: Humoral Immune Response for Each Vaccine Strain in Terms of Haemagglutination Inhibition (HI) Antibody Titers.
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Switzerland/9715293/2013 (H3N2), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Days 0 and 21.
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available and subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 62 | 57
Titers
  H1N1, Day 0 | 47.3 [32.2 to 69.4] | 31.2 [22.6 to 42.9]
  H1N1, Day 21 | 460.2 [346.7 to 610.8] | 166.9 [125.6 to 221.9]
  H3N2, Day 0 | 32.0 [22.6 to 45.3] | 41.7 [29.0 to 60.0]
  H3N2, Day 21 | 338.4 [257.3 to 445.0] | 306.7 [224.5 to 418.9]
  Yamagata, Day 0 | 84.1 [58.4 to 121.0] | 77.6 [62.2 to 96.8]
  Yamagata, Day 21 | 338.4 [266.7 to 429.3] | 226.3 [184.6 to 277.3]
  Victoria, Day 0 | 68.8 [51.3 to 92.2] | 99.6 [74.2 to 133.6]
  Victoria, Day 21 | 365.9 [291.3 to 459.5] | 288.6 [223.7 to 372.3]

2. Primary Outcome: Number of Seropositive Subjects for HI Antibodies Against Each of the 4 Vaccine Strains.
Description: A seropositive subject was a subject whose HI antibody titer was greater than or equal to the assay cutoff value of 1:10. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Switzerland/9715293/2013 (H3N2), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 62 | 57
Subjects
  H1N1, Day 0 | 51 | 52
  H1N1, Day 21 | 62 | 57
  H3N2, Day 0 | 52 | 52
  H3N2, Day 21 | 62 | 57
  Yamagata, Day 0 | 59 | 57
  Yamagata, Day 21 | 62 | 57
  Victoria, Day 0 | 59 | 57
  Victoria, Day 21 | 62 | 57

3. Primary Outcome: Number of Subjects Who Were Seroprotected for Anti-HI Antibodies Against Each of the 4 Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Switzerland/9715293/2013 (H3N2), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 62 | 57
Subjects
  H1N1, Day 0 | 40 | 31
  H1N1, Day 21 | 62 | 54
  H3N2, Day 0 | 29 | 33
  H3N2, Day 21 | 61 | 55
  Yamagata, Day 0 | 46 | 47
  Yamagata, Day 21 | 62 | 57
  Victoria, Day 0 | 48 | 48
  Victoria, Day 21 | 62 | 57

4. Primary Outcome: Number of Seroconverted Subjects for Anti-HA Antibodies Against Each of the 4 Vaccine Influenza Strains.
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination HI titer less than (<) 1:10 and a post-vaccination HI titer ≥1:40 or pre-vaccination HI titer ≥ 1:10 and at least a 4-fold increase in post-vaccination HI titer. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Switzerland/9715293/2013 (H3N2), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Day 21.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 62 | 57
Subjects
  H1N1 | 38 | 35
  H3N2 | 49 | 41
  Yamagata | 31 | 20
  Victoria | 38 | 20

5. Primary Outcome: Number of Subjects With Seroprotection Power (SPP) for HI Antibody Titer Against Each of the 4 Vaccine Influenza Strains Above the Cut-off Value.
Description: SPP was defined as the number of vaccinated subjects with a pre-vaccination titer < 1:40 and a post-vaccination titer ≥ 1:40.
  The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Switzerland/9715293/2013 (H3N2), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 62 | 57
Subjects
  H1N1 | 22 | 23
  H3N2 | 32 | 22
  Yamagata | 16 | 10
  Victoria | 14 | 9

6. Primary Outcome: Mean Geometric Increase (MGI) for HI Antibody Titer Against Each of the 4 Vaccine Influenza Strains.
Description: MGI also known as the seroconversion factor [SCF] was defined as the fold increase in serum HI GMTs post vaccination compared to pre-vaccination (Day 0). The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Switzerland/9715293/2013 (H3N2), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 62 | 57
Fold increase
  H1N1 | 9.7 [5.9 to 16.1] | 5.4 [3.8 to 7.5]
  H3N2 | 10.6 [7.7 to 14.6] | 7.4 [5.3 to 10.2]
  Yamagata | 4.0 [3.0 to 5.4] | 2.9 [2.3 to 3.7]
  Victoria | 5.3 [3.8 to 7.5] | 2.9 [2.2 to 3.9]

7. Secondary Outcome: Humoral Immune Response for Each Vaccine Strain in Terms of HI Antibodies.
Description: Antibody titers were expressed as GMTs. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Switzerland/9715293/2013 (H3N2), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Fluarix Tetra (Southern Hemisphere) Adult Group_Y: Subjects aged 18-60 years administered with the study vaccine [1 dose of Fluarix™ Tetra (Southern Hemisphere) vaccine at Day 0, administered intramuscularly in the deltoid of the non-dominant arm] and who had received vaccination in 2014.
- Fluarix Tetra (Southern Hemisphere) Adult Group_N: Subjects aged 18-60 years administered with the study vaccine [1 dose of Fluarix™ Tetra (Southern Hemisphere) vaccine at Day 0, administered intramuscularly in the deltoid of the non-dominant arm] and who had not received vaccination in 2014.
- Fluarix Tetra (Southern Hemisphere) Elderly Group_Y: Subjects aged >60 years administered with the study vaccine [1 dose of Fluarix™ Tetra (Southern Hemisphere) vaccine at Day 0, administered intramuscularly in the deltoid of the non-dominant arm] and who had received vaccination in 2014.
- Fluarix Tetra (Southern Hemisphere) Elderly Group_N: Subjects aged >60 years administered with the study vaccine [1 dose of Fluarix™ Tetra (Southern Hemisphere) vaccine at Day 0, administered intramuscularly in the deltoid of the non-dominant arm] and who had not received vaccination in 2014.
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group_Y | Fluarix Tetra (Southern Hemisphere) Adult Group_N | Fluarix Tetra (Southern Hemisphere) Elderly Group_Y | Fluarix Tetra (Southern Hemisphere) Elderly Group_N
Number analyzed (Participants) | 31 | 31 | 46 | 11
Titers
  H1N1, Day 0 | 86.5 [56.7 to 132.0] | 25.9 [14.4 to 46.5] | 33.9 [23.4 to 48.9] | 22.0 [11.0 to 43.9]
  H1N1, Day 21 | 276.7 [206.8 to 370.3] | 765.3 [499.0 to 1174.0] | 151.8 [111.2 to 207.0] | 248.7 [115.6 to 534.9]
  H3N2, Day 0 | 41.3 [26.1 to 65.5] | 24.7 [14.5 to 42.2] | 44.8 [30.1 to 66.5] | 31.0 [11.1 to 87.1]
  H3N2, Day 21 | 342.2 [240.9 to 486.1] | 334.6 [215.2 to 520.3] | 281.6 [196.3 to 403.9] | 438.5 [229.9 to 836.4]
  Yamagata, Day 0 | 133.7 [89.2 to 200.4] | 52.9 [29.5 to 94.6] | 88.2 [70.2 to 110.8] | 45.4 [24.7 to 83.5]
  Yamagata, Day 21 | 306.0 [223.4 to 419.0] | 374.2 [257.8 to 543.1] | 194.6 [157.6 to 240.3] | 425.0 [267.3 to 675.7]
  Victoria, Day 0 | 95.6 [68.7 to 133.0] | 49.5 [30.7 to 79.6] | 114.9 [82.7 to 159.5] | 54.8 [29.3 to 102.8]
  Victoria, Day 21 | 282.9 [207.7 to 385.3] | 473.2 [341.5 to 655.7] | 259.2 [196.3 to 342.3] | 452.5 [236.2 to 867.1]

8. Secondary Outcome: Number of Seropositive Subjects for HI Antibodies Against Each of the 4 Vaccine Strains.
Description: as for outcome 2
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group_Y | Fluarix Tetra (Southern Hemisphere) Adult Group_N | Fluarix Tetra (Southern Hemisphere) Elderly Group_Y | Fluarix Tetra (Southern Hemisphere) Elderly Group_N
Number analyzed (Participants) | 31 | 31 | 46 | 11
Subjects
  H1N1, Day 0 | 30 | 21 | 42 | 10
  H1N1, Day 21 | 31 | 31 | 46 | 11
  H3N2, Day 0 | 30 | 22 | 43 | 9
  H3N2, Day 21 | 31 | 31 | 46 | 11
  Yamagata, Day 0 | 31 | 28 | 46 | 11
  Yamagata, Day 21 | 31 | 31 | 46 | 11
  Victoria, Day 0 | 31 | 28 | 46 | 11
  Victoria, Day 21 | 31 | 31 | 46 | 11

9. Secondary Outcome: Number of Subjects Who Were Seroprotected for Anti-HI Antibodies Against Each of the 4 Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer ≥ 1:40 that usually is accepted as indicating protection in adults. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Switzerland/9715293/2013 (H3N2), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group_Y | Fluarix Tetra (Southern Hemisphere) Adult Group_N | Fluarix Tetra (Southern Hemisphere) Elderly Group_Y | Fluarix Tetra (Southern Hemisphere) Elderly Group_N
Number analyzed (Participants) | 31 | 31 | 46 | 11
Subjects
  H1N1, Day 0 | 27 | 13 | 27 | 4
  H1N1, Day 21 | 31 | 31 | 43 | 11
  H3N2, Day 0 | 16 | 13 | 28 | 5
  H3N2, Day 21 | 31 | 30 | 44 | 11
  Yamagata, Day 0 | 28 | 18 | 41 | 6
  Yamagata, Day 21 | 31 | 31 | 46 | 11
  Victoria, Day 0 | 27 | 21 | 41 | 7
  Victoria, Day 21 | 31 | 31 | 46 | 11

10. Secondary Outcome: MGI for HI Antibody Titer Against Each of the 4 Vaccine Influenza Strains.
Description: as for outcome 6
Time Frame: At Day 21
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group_Y | Fluarix Tetra (Southern Hemisphere) Adult Group_N | Fluarix Tetra (Southern Hemisphere) Elderly Group_Y | Fluarix Tetra (Southern Hemisphere) Elderly Group_N
Number analyzed (Participants) | 31 | 31 | 46 | 11
Fold increase
  H1N1 | 3.2 [2.3 to 4.5] | 29.6 [13.5 to 64.8] | 4.5 [3.2 to 6.3] | 11.3 [4.1 to 31.1]
  H3N2 | 8.3 [5.4 to 12.7] | 13.5 [8.3 to 22.2] | 6.3 [4.5 to 8.8] | 14.1 [4.9 to 40.8]
  Yamagata | 2.3 [1.7 to 3.0] | 7.1 [4.4 to 11.3] | 2.2 [1.8 to 2.6] | 9.4 [4.2 to 21.0]
  Victoria | 3.0 [2.1 to 4.1] | 9.6 [5.6 to 16.4] | 2.3 [1.8 to 2.9] | 8.3 [3.1 to 21.9]

11. Secondary Outcome: Number of Seroconverted Subjects for Anti-HA Antibodies Against Each of the 4 Vaccine Influenza Strains.
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination HI titer less than (<) 1:10 and a post-vaccination HI titer ≥1:40 or pre-vaccination HI titer ≥1:10 and at least a 4-fold increase in post-vaccination HI titer. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Switzerland/9715293/2013 (H3N2), Flu B/Phuket/3073/2013 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Day 21.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group_Y | Fluarix Tetra (Southern Hemisphere) Adult Group_N | Fluarix Tetra (Southern Hemisphere) Elderly Group_Y | Fluarix Tetra (Southern Hemisphere) Elderly Group_N
Number analyzed (Participants) | 31 | 31 | 46 | 11
Subjects
  H1N1 | 14 | 24 | 26 | 9
  H3N2 | 25 | 24 | 33 | 8
  Yamagata | 8 | 23 | 12 | 8
  Victoria | 14 | 24 | 13 | 7

12. Secondary Outcome: Number of Subjects With Seroprotection Power (SPP) for HI Antibody Titer Against Each of the 4 Vaccine Influenza Strains Above the Cut-off Value.
Description: as for outcome 5
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group_Y | Fluarix Tetra (Southern Hemisphere) Adult Group_N | Fluarix Tetra (Southern Hemisphere) Elderly Group_Y | Fluarix Tetra (Southern Hemisphere) Elderly Group_N
Number analyzed (Participants) | 31 | 31 | 46 | 11
Subjects
  H1N1 | 4 | 18 | 16 | 7
  H3N2 | 15 | 17 | 16 | 6
  Yamagata | 3 | 13 | 5 | 5
  Victoria | 4 | 10 | 5 | 4

13. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as pain that prevented normal everyday activities. Grade 3 redness and swelling was greater than 100 millimeters (mm) i.e. >100mm.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: Analysis was performed on the Total Vaccinated cohort, which included all subjects with vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 62 | 57
Subjects
  Any Pain | 27 | 13
  Grade 3 Pain | 3 | 0
  Any Redness | 9 | 7
  Grade 3 Redness | 0 | 0
  Any Swelling | 7 | 6
  Grade 3 Swelling | 0 | 0

14. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were Arthralgia, Fatigue, Gastrointestinal symptoms, Headache, Myalgia, Shivering, Sweating and Temperature (Oral). Any was defined as any general symptom reported irrespective of intensity or relationship to vaccination. Grade 3 was defined as symptoms that prevented normal activity. Related was defined as general symptom assessed by the investigator to have a causal relationship to vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 13
Measure: Number; unit: Subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 62 | 57
Subjects
  Any Arthralgia | 6 | 2
  Grade 3 Arthralgia | 0 | 1
  Related Arthralgia | 5 | 1
  Any Fatigue | 6 | 1
  Grade 3 Fatigue | 1 | 0
  Related Fatigue | 5 | 0
  Any Gastrointestinal symptoms | 3 | 0
  Grade 3 Gastrointestinal symptoms | 0 | 0
  Related Gastrointestinal symptoms | 2 | 0
  Any Headache | 8 | 1
  Grade 3 Headache | 2 | 1
  Related Headache | 6 | 1
  Any Myalgia | 9 | 2
  Grade 3 Myalgia | 0 | 1
  Related Myalgia | 8 | 1
  Any Sweating | 2 | 0
  Grade 3 Sweating | 1 | 0
  Related Sweating | 2 | 0
  Any Shivering | 2 | 0
  Grade 3 Shivering | 0 | 0
  Related Shivering | 1 | 0
  Any Temperature (Oral) | 0 | 0
  Grade 3 Temperature (Oral) | 0 | 0
  Related Temperature (Oral) | 0 | 0

15. Secondary Outcome: Duration of Solicited Local Symptoms
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 13
Measure: Median (Full Range); unit: days
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 27 | 13
days
  Pain (N = 27, 13) | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 3.0]
  Redness (N = 9, 7) | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0]
  Swelling (N = 7, 6) | 3.0 [1.0 to 4.0] | 1.5 [1.0 to 2.0]

16. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Medically Attended Adverse Events (MAEs).
Description: MAEs were defined as AEs with a medically-attended visit i.e. prompting emergency room (ER) visits, hospitalizations or physician visits and that were not routine visits for physical examination or vaccination. Any MAE was defined as at least one MAE experienced. Grade 3 was defined as MAEs that prevented normal activities and related was defined as MAEs assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the entire study period (approximately 21 days for each subject).
Population: as for outcome 13
Measure: Number; unit: subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 63 | 57
subjects
  Any MAEs | 4 | 6
  Grade 3 MAEs | 3 | 1
  Related MAEs | 0 | 0

17. Secondary Outcome: Duration of Solicited General Symptoms
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 13
Measure: Median (Full Range); unit: days
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 9 | 2
days
  Arthralgia [N = 6,2] | 1.5 [1.0 to 3.0] | 2.5 [1.0 to 4.0]
  Fatigue [N = 6,1] | 3.0 [1.0 to 4.0] | 2.0 [2.0 to 2.0]
  Gastrointestinal symptoms [N = 3,0] | 1.0 [1.0 to 3.0] | 0.0 [0.0 to 0.0]
  Headache [N = 8,1] | 2.5 [1.0 to 3.0] | 1.0 [1.0 to 1.0]
  Myalgia [N = 9,2] | 2.0 [1.0 to 4.0] | 3.0 [2.0 to 4.0]
  Sweating [N = 2,0] | 2.5 [1.0 to 4.0] | 0.0 [0.0 to 0.0]
  Shivering [N = 2,0] | 1.5 [1.0 to 2.0] | 0.0 [0.0 to 0.0]

18. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was an event that prevented normal activities and related was defined as an unsolicited AE assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the 21-day (Days 0-20) post-vaccination period.
Population: as for outcome 13
Measure: Number; unit: Subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 63 | 57
Subjects
  Any Unsolicted AEs | 11 | 10
  Grade 3 Unsolicted AEs | 4 | 2
  Related Unsolicted AEs | 4 | 0

19. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: A serious adverse event was any untoward medical occurrence that: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (approximately 21 days for each subject)
Population: as for outcome 13
Measure: Number; unit: Subjects
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Number analyzed (Participants) | 63 | 57
Subjects
  Any SAEs | 0 | 1
  Related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse events (SAE) =Entire study period. Solicited local and general symptoms = During the 4-day follow up period post vaccination. Unsolicited AEs = during the 21-day follow-up period after vaccination.
Groups:
- Fluarix Tetra (Southern Hemisphere) Elderly Group: Subjects aged ˃60 years received 1 dose of Fluarix™ Tetra (Southern Hemisphere) vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
Arm/Group | Fluarix Tetra (Southern Hemisphere) Adult Group | Fluarix Tetra (Southern Hemisphere) Elderly Group
Serious Adverse Events (participants affected / at risk) | 0/63 | 1/57
Other Adverse Events (participants affected / at risk) | 27/63 | 13/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluarix Tetra (Southern Hemisphere) Adult Group (N=63) | Fluarix Tetra (Southern Hemisphere) Elderly Group (N=57)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluarix Tetra (Southern Hemisphere) Adult Group (N=63) | Fluarix Tetra (Southern Hemisphere) Elderly Group (N=57)
Fatigue (General disorders) | 6 (6) | 2 (2)
Pain (General disorders) | 27 (27) | 13 (13)
Swelling (General disorders) | 7 (7) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 3 (3)
Headache (Nervous system disorders) | 8 (8) | 1 (1)
Erythema (redness) (Skin and subcutaneous tissue disorders) | 9 (9) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.